CLINICAL TRIAL: NCT03880825
Title: A Phase I Open-Label, Fixed-Sequence Pharmacokinetic Drug Interaction Study to Evaluate the Effect of Levoketoconazole on the Single-Dose Pharmacokinetics of Metformin in Healthy Subjects
Brief Title: Drug Interaction Study of Levoketoconazole and Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortendo AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: COR-2017-03
Record Dates: First submitted 2019-03-18; First posted 2019-03-19 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Metformin; Tablets; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Metformin Only (Other)
  Interventions: Drug: Metformin 500 mg Oral Tablet
- Levoketoconazole Only (Other)
  Interventions: Drug: Levoketoconazole 150 - 600 mg (BID)
- Levoketoconazole + Metformin (Other)
  Interventions: Drug: Metformin 500 mg Oral Tablet; Drug: Levoketoconazole 150 - 600 mg (BID)

INTERVENTIONS:
Drug: Metformin 500 mg Oral Tablet — single dose
  Arms: Levoketoconazole + Metformin; Metformin Only
Drug: Levoketoconazole 150 - 600 mg (BID) — escalating dose from 150 mg to 600 mg (BID)
  Other Names: COR-003
  Arms: Levoketoconazole + Metformin; Levoketoconazole Only

SUMMARY:
This is a phase I, open-label, fixed-sequence drug-drug interaction study to evaluate the effect of levoketoconazole on the single-dose PK of metformin in health subjects.

DETAILED DESCRIPTION:
This study will enroll healthy male and female subjects to evaluate the effect of levoketoconazole on the PK of a single 500 mg dose of metformin. There will be 3 sequential treatment periods, and all subjects will receive metformin only in Period 1, escalating doses of levoketoconazole in Period 2, and concurrent administration of metformin and levoketoconazole in Period 3.

ELIGIBILITY:
Inclusion Criteria:

1. 18-55 years of age, inclusive, at time of consent.
2. Body mass index (BMI) between 18 and 32 kg/m2, inclusive.
3. In good general physical health as determined by absence of clinically significant medical history, physical examination findings, vital signs, clinical laboratory evaluations and ECG measurements.
4. Has not consumed and agrees to abstain from taking any prescription drugs, dietary supplements including vitamins and herbal preparations, or non-prescription drugs (except as authorized by the Investigator AND Medical Monitor) for 14 days prior to initial CRU admission on Day -1 and through Follow-Up.
5. Has not consumed alcohol-containing beverages for 3 days prior to initial CRU admission on Day -1 and agrees not to consume alcohol for the duration of the study through Follow-Up.
6. Is a nonsmoker (for at least 3 months) with negative urinary cotinine test at Screening and agrees to abstain from tobacco- and nicotine containing products for the duration of the study.

Exclusion Criteria:

1. Evidence of any out-of-normal-range laboratory value at Screening that has not been reviewed, approved, and documented as Not Clinically Significant by the Investigator (except for LFTs, which must be within the normal range).
2. Concurrent medical illness that would interfere with the conduct of the study in the opinion of the Investigator.
3. History or presence of clinically significant cardiovascular, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, psychiatric, renal, hepatic, chronic respiratory, or gastrointestinal disease as judged by the Investigator.
4. Clinically significant ECG abnormality or confirmed QTcF interval > 450 msec at Screening or unconfirmed QTcF interval > 450 msec at CRU admission.
5. Family history (parents, siblings, and offspring) of QT interval sudden cardiac death.
6. Positive urine drug screen for drugs-of-abuse, including cocaine, 3,4 methylenedioxy-methamphetamine (MDMA), tetrahydrocannabinol, opioids, benzodiazepines, amphetamines, and barbiturates, and/or positive urine screen for alcohol at Screening and CRU admission.
7. Positive urinary cotinine test at Screening.
8. Treatment with an investigational drug within the longer of 30 days or five half-lives of the investigational drug preceding the first dose of study drug.
9. Positive for Human Immunodeficiency Virus (HIV), hepatitis B, and/or hepatitis C on Screening assessments.
10. Acute illness within 7 days of the first CRU admission on Day -1.
11. Donated plasma within 7 days of Screening.
12. Donated 1 or more pints of blood (or equivalent blood loss) within 30 days prior to Screening.
13. History of caffeine consumption exceeding 8 cups of coffee/day (1 cup = 8 fluid ounces) within 14 days prior to first dose, or consumption of any caffeine- or chocolate-containing products for 3 days prior to CRU admission each week. Caffeine containing foods and/or beverages (e.g., tea and cola) should be considered equivalent to coffee.
14. History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of hard liquor) within 180 days of Screening.
15. Female subject who is pregnant or lactating.
16. Male with hemoglobin less than 12.0 g/dL; Female with hemoglobin less than 11.0 g/dL.
17. Had difficulties swallowing whole tablets.
18. Body habitus prevents repeated venipuncture.
19. History of hypersensitivity or allergy to metformin.
20. History of hypoglycemia.
21. Participated in the COR-2017-02 levoketoconazole food effect study.
22. History of drug-induced liver injury from any drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of metformin | 48 hours
  Maximum observed plasma concentration (Cmax) of metformin with and without concomitant administration of levoketoconazole.
Time to maximum concentration (Tmax) of metformin | 48 hours
  Time to maximum concentration (Tmax) of metformin with and without concomitant administration of levoketoconazole.
Area under the plasma concentration-time curve (AUC) of metformin | 48 hours
  Area under the plasma concentration-time curve (AUC) from time 0 to time of last measurable plasma concentration (AUClast) and from time 0 extrapolated to infinity (AUCinf) of metformin with and without concomitant administration of levoketoconazole.

SECONDARY OUTCOMES:
Renal clearance (CLr) of metformin | 24 hours
  Renal clearance (CLr) of metformin with and without concomitant administration of levoketoconazole.
Incidence of Adverse Events | 35 days
  Incidence of Treatment-Emergent AEs (TEAEs), AESIs, and Serious Adverse Events (SAEs).
  Incidence of Treatment-Emergent AEs (TEAEs), AESIs, and Serious Adverse Events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Schoenfeld, MD, Study Director — Cortendo AB
Locations (1):
- Clinical Pharmacology of Miami, LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No